CLINICAL TRIAL: NCT00821652
Title: Phase I Randomized, Double-blind, Placebo-controlled Study of Topical Resiquimod as an Adjuvant for NY-ESO1 Protein+Montanide Vaccination in Patients With Tumors That Often Express NY-ESO-1
Brief Title: Randomized, Double Blind, Placebo-controlled Topical Resiquimod Adjuvant for NY-ESO-1 Protein Vaccination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nina Bhardwaj (Other)
Collaborators: Cancer Research Institute, New York City (Other)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Director, Immunotherapy Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 13-1390
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Tumors
Keywords: Tumor; NY-ESO-1 expression; Tumors that often express NY-ESO-1.
MeSH Terms: conditions — Neoplasms | interventions — resiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose-esclation (Other): Part I represents a dose-escalation part with topical resiquimod in an open-label fashion.
  Interventions: Drug: NY-ESO-1 protein; Montanide ISA®-51 VG; Resiquimod
- 2 (Experimental): Part II: Eligible patients will be randomized to receive a subcutaneous vaccination of 100µg NY-ESO-1 protein emulsified in 1.25mL Montanide ISA®-51 VG (day 1) followed by topical placebo gel (Arm A) or topical resiquimod gel (Arm B) on days 1, 3 and 5; or resiquimod dosing regimen established in Part I.
  Interventions: Drug: NY-ESO-1 protein; Montanide ISA®-51 VG; Resiquimod/placebo

INTERVENTIONS:
Drug: NY-ESO-1 protein; Montanide ISA®-51 VG; Resiquimod — Part I: a cohort of 3 patients to receive a subcutaneous vaccination of 100µg NY-ESO-1 protein emulsified in 1.25mL Montanide ISA®-51 VG (day 1) followed by topical resiquimod 1000 mg of the 0.2% gel on days 1, and 3. If no DLT observed, we will proceed to cohort 2 with Resiquimod dosing on days 1,3 and 5. If DLT is found in the second cohort, the trial will proceed to Part II; with the limited dosing for days 1 and 3 only, as used in the first cohort. If no DLT is found in second cohort, the trial will proceed to Part II with Resiquimod dosing for days1, 3 and 5.
  Arms: Dose-esclation
Drug: NY-ESO-1 protein; Montanide ISA®-51 VG; Resiquimod/placebo — Part II: Eligible patients will be randomized to receive a subcutaneous vaccination of 100µg NY-ESO-1 protein emulsified in 1.25mL Montanide ISA®-51 VG (day 1) followed by topical placebo gel (Arm A) or topical resiquimod gel (Arm B) on days 1, 3 and 5; or resiquimod dosing regimen established in Part I. The cycles will be repeated every 3 weeks for a total of 4 cycles (on Study week 1, 4, 7 and 10). All procedures may occur within + 3 days of the planned date.
  Arms: 2

SUMMARY:
The study is designed to see if a course of injections containing the NY-ESO-1 protein (a tumor antigen, marker expressed by tumors); in combination with an immune stimulant (adjuvant) Montanide, with or without resiquimod (another adjuvant) is well tolerated and safe in patients with surgically resected Stage IIB, IIC, Stage III or Stage IV (AJCC criteria) melanoma, a tumor that expresses NY-ESO-1. In addition, this study is designed to see if the patient's body's defense (immune) system can be boosted (strengthened) by this vaccine and if the addition of resiquimod to the vaccine makes this more likely.

DETAILED DESCRIPTION:
There is no published data on the application of topical resiquimod in combination with an antigen in Montanide, therefore, this study includes a 2-part design where Part I represents a dose-escalation part with topical resiquimod in an open-label fashion. Part II represents the randomized part.

In Part I, 2 cohorts are planned: If no dose-limiting toxicity (DLT) occurs by day 8 of the last vaccination cycle in the last patient enrolled the first cohort, 3 additional patients (cohort 2) will be enrolled. If no DLT occurs by day 8 of the last vaccination cycle in the last patient enrolled the second cohort in Part I, the trial will proceed to Part II where patients will be randomized.

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible for enrollment if they fulfill the following criteria:

1. Histological diagnosis of surgically resected Stage IIB, IIC, Stage III or Stage IV (AJCC criteria) melanoma independent of NY-ESO-1 expression in a tumor biopsy
2. At least 4 weeks since surgery prior to first dosing of study agent.
3. Laboratory values within the following limits:

   Hemoglobin > 10.0 g/dL Neutrophil count > 1.5 x l09/L Lymphocyte count > Lower limit of institutional normal Platelet count > 80 x l09/L Serum creatinine < 2.0 mg/dL Serum bilirubin < 2 x upper limit of institutional normal AST/ALT < 2 x upper limit of institutional normal
4. Patients must have an ECOG performance status of <2 (ECOG criteria published in [46])
5. Life expectancy > 6 months.
6. Age > 18 years.
7. Able and willing to give written informed consent for participation in the trial (see Section 12.2)
8. Patients enrolled in the adjuvant setting must have received standard curative therapy, e.g., surgery, radiation. Alternatively, patients can enter after refusing standard curative therapy only if therapy was clearly discussed with the treating physician or if they have failed another biologic therapy due to toxicity.

Exclusion Criteria

Patients will be excluded from the study if they fulfill any of the following criteria:

1. Serious illnesses, e.g., serious infections requiring antibiotics.
2. Previous bone marrow or stem cell transplant.
3. History of immunodeficiency disease (such as HIV) or autoimmune disease except vitiligo.
4. Metastatic disease to the central nervous system.
5. Other malignancy prior to entry into the study.
6. No radiation therapy, prior biological therapy or surgery within 4 weeks prior to first dose of study agent.
7. No prior chemotherapy or prior vaccine or immunotherapy.
8. Concomitant treatment with systemic corticosteroids greater than physiologic doses. Topical (but not at the proposed vaccination sites) or inhalational steroids are permitted. (See also Section 6.7 for restrictions/recommendations on 'Ancillary Therapy'.)
9. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent.
10. Pregnancy or lactation.
11. Women of childbearing potential not using a medically acceptable means of contraception.
12. Patients with known history of inflammatory skin disorders (e.g.,psoriasis, lupus) that may be exacerbated by Resiquimod.
13. Psychiatric or addictive disorders that may compromise the ability to give informed consent.
14. Lack of availability of the patient for immunological and clinical follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary objectives of the study are to define the safety and immunogenicity of vaccination with NY-ESO-1 protein emulsified in Montanide® ISA-51 VG when given with or without the topical TLR 7/8 agonist resiquimod. | Blood samples are obtained at baseline, 1 week after each vaccination, and at follow-up 1visit.

SECONDARY OUTCOMES:
To document tumor response by RECIST criteria if applicable. Skin section analysis of resiquimod/placebo treated site for immune cell infiltration and gene expression analysis. Investigation of polymorphisms for TLR7/8 through germline SNP analysis | Skin biopsies will be obtained after the last vaccination cycle. Clinical hematology and biochemistry measurements will be taken at baseline, one week after the second vaccination and two to four weeks after the fourth vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Rachel Sabado, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States